CLINICAL TRIAL: NCT06762366
Title: Substitution in Adult Proportional Reasoning
Brief Title: Substitution Heuristic on Proportional Tasks
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Hurst, PhD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor-Investigator, Michelle Hurst, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2024002168; R00HD104990 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Proportional Reasoning; Substitution Heuristic
Keywords: proportion; hueristic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Additional Incentive (Active Comparator): In this arm of the experiment, participants will receive the additional incentive intervention.
  Interventions: Behavioral: Additional Incentive
- Response Delay (Active Comparator): In this arm of the experiment, participants will receive the response delay intervention.
  Interventions: Behavioral: Response Delay
- Baseline Performance (Sham Comparator): In this arm of the study, participants will complete the task as it is typically administed.
  Interventions: Behavioral: Baseline Performance

INTERVENTIONS:
Behavioral: Additional Incentive — During this behavioral intervention, participants will be given additional compensation for correct answers.
  Arms: Additional Incentive
Behavioral: Response Delay — During this behavioral intervention, participants will not be allowed to respond with their judgements until after a certain amount of time has passed.
  Arms: Response Delay
Behavioral: Baseline Performance — In this intervention, the participant completes the task as it is typically administer for a baseline performance measure. The participant can respond at will and does not receive incentive for correct responses.
  Arms: Baseline Performance

SUMMARY:
The goal of this clinical trial is to test whether or not adults use a substitution heuristic when reasoning about proportions. The main question it aims to answer is:

Do adults use a substitution heuristic when judging non-symbolic proportions, leading them to answer an easier, yet incorrect question?

Researchers will compare performance at baseline with one of two conditions in order to see if forced behavioral changes can change performance on the task.

Participants will be asked to compare two images and judge which has the higher proportion of the target color. Each participant will also be assigned to one of two condition where they either receive a further incentive for correct selections or are required to use more time when making their calculations.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing people within the target age range

Exclusion Criteria:

* Individuals with known developmental or cognitive disorders
* Participants must speak/read sufficient English to read and complete the informed consent document

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Proportion Correct | up to 20 minutes
  Accuracy will be measured for each trial and combined into an overall score (i.e., proportion of trials correct).
Reaction Time | up to 20 minutes
  Reaction time will also be tracked (i.e., time it takes to respond), with a faster reaction time indicating ease and/or efficiency with the task.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Center for Cognitive Science, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participant responses to all measures, as well as de-identified demographics (e.g., age, gender) will be made publicly available on a data repository.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning when the results are published (if not earlier) with no planned end date.
Access Criteria: De-identified data will be publicly available under a creative commons license only requesting attribution.

DOCUMENTS (1):
  • Informed Consent Form (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT06762366/ICF_000.pdf